CLINICAL TRIAL: NCT01308073
Title: Long-time Stability of Middle Molecule Clearance During CI-Ca CVVHD
Brief Title: Stability of Middle Molecule Clearance
Acronym: EMIC2
Status: Completed | Type: Observational
Sponsor: Klinik für Anästhesiologie (Other)
Collaborators: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor-Investigator, Klinik für Anästhesiologie, Leiter Interdisziplinäre Operative Intensivstation ZOM-I, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Other Study IDs: EMIC2_2011_02_03
Record Dates: First submitted 2011-02-04; First posted 2011-03-03 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Continuous Hemodialysis
MeSH Terms: interventions — Renal Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EMIC 2 dialysis: Patients on ICU requiring dialysis for acute renal insufficiency
  Interventions: Device: Hemodialysis with EMIC 2 filters

INTERVENTIONS:
Device: Hemodialysis with EMIC 2 filters — Patients with indication for routine continuous hemodialysis due to acute renal insufficiency

SUMMARY:
The investigators aim to show, whether all middle molecules are included in the clearance and whether this clearance is stable until 72 hours.

DETAILED DESCRIPTION:
A better middle molecule clearance has been shown until 24 hours of duration. The investigators will extend our observations until 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age>18 years
* acute renal insufficiency with indication for continuous hemodialysis, according to RILFE classification F: serum creatinine increase > 3-fold or serum creatinine > 4mg/dl with acute increase of >0,5mg/dl Urine Output <0,3mg/kg/h for 24 h or anuria for 12 h
* body weight:60-80kg
* anticoagulation with citrate possible and indicated
* Dose for hemodialysis of 2l/h

Exclusion Criteria:

* participation in another clinical trial within on month prior to this study
* pregnancy or brest feeding
* septic shock
* interference with cystatin-C

  1. haemolysis <1g/dl
  2. Bilirubin<9mg/dl
  3. Triglyceride >700mg/dl
  4. rheumatoid factor > 300kIU/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of surgical intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Clearance of Urea | up to 72 h
Clearance of Cystatin C | up to 72 h
Clearance of creatinine | up to 72 h
Clearance of Beta2-Microglobulin | up to 72 h
Clearance of Osteocalcin | up to 72 h
Free light chains kappa of Immunoglobulins | up to 72 h
Clearance of albumin | up to 72 h

SECONDARY OUTCOMES:
Mean arterial pressure | up to 72 h
Vasopressor requirement | up to 72 h
Heart rate | up to 72 h

CONTACTS AND LOCATIONS:
Overall Officials: Detlef Kindgen-Milles, Prof., Principal Investigator — Klinik für Anästhesiologie Universitätsklinikum Düsseldorf Heinrich-Heine Universität
Locations (1):
- Intensivstation ZOM1 Klinik für Anästhesiologie Universitätsklinikum Düsseldorf, Düsseldorf, Germany